CLINICAL TRIAL: NCT03026361
Title: Molecular Mechanisms of Precancerous and Cancerous Lesions of the Oral Cavity
Brief Title: Molecular Mechanisms of the Development of Precancerous and Cancerous Lesions of the Oral Cavity
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Principal Investigator, Marinka Mravak Stipetic, Professor, University of Zagreb
Other Study IDs: 06509824642532
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Oral Lichen Planus; Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Lichen Planus, Oral; Squamous Cell Carcinoma of Head and Neck | interventions — Immunohistochemistry; Blotting, Western

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- oral lichen planus (OLP): Histopathologically confirmed samples of OLP underwent immunohistochemical analysis of IGF2 and IGF2R expression.
  Fresh-frozen samples of clinically OLP changed and adjacent healthy mucosa underwent global proteomic profiling and two proteins were subsequently validated with Western blot.
  Interventions: Genetic: global proteomic profiling
- oral squamous cell carcinoma (OSCC): Histopathologically confirmed samples of OSCC underwent immunohistochemical analysis of IGF2 and IGF2R expression.
  Fresh-frozen samples of clinically OSCC changed and adjacent healthy mucosa underwent global proteomic profiling and two proteins were subsequently validated with Western blot.
  Interventions: Genetic: global proteomic profiling
- healthy mucosa: Archival samples of healthy oral mucosa underwent immunohistochemical analysis of IGF2 and IGF2R expression.
  Fresh-frozen samples of healthy mucosa taken during alveolotomy underwent global proteomic profiling and two proteins were subsequently validated with Western blot.
  Interventions: Genetic: global proteomic profiling

INTERVENTIONS:
Genetic: global proteomic profiling — Global proteomic profiling was performed on OLP and OSCC samples and healthy mucosa. Obtained data was analysed in Uniprot database (http://uniprot.org) with the emphasis on extracellular matrix proteins. In total, 55 extracellular matrix proteins were found to be expressed in analysed samples with very high confidence.
  Other Names: immunohistochemistry; Western blot

SUMMARY:
The aim of this study was to examine molecular alterations on the protein level in lesions of oral lichen planus (OLP), oral squamous cell carcinoma (OSCC) and healthy mucosa. Global protein profiling methods based on liquid chromatography coupled to mass spectrometry were used, with a special emphasis on evaluation of deregulated extracellular matrix molecules expression, as well as on analyses of insulin-like growtg factor 2 (IG2F) and insulin-like growth factor 2 receptor (IGFR2) expression in healthy mucosa, OLP and OSCC tissues by comparative semiquantitative immunohistochemistry.

Mass spectrometry based proteomics profiling of healthy mucosa, OLP and OSCC tissues (and accompanied histologically unaltered tissues, respectively) identified 55 extracellular matrix proteins. Twenty among identified proteins were common to all groups of samples. Statistically significant difference between final IGF2 and IGF2R IRS scores in favour to IGF2R may further corroborate the IG2FR antitumor role in OLP and OSCC where it acts as a negative regulator of IGF2 activity.

DETAILED DESCRIPTION:
Although OLP is categorised as a precancerous condition associated with a significantly increased risk of oral cancer, molecular pathophysiology of OLP and its potential for malignant transformation in OSCC are poorly understood and remain controversial. Development of new analytical methods enhances research in the field of malignant disorders. Identification of novel biomarkers help in the diagnostic process, pre-symptomatic interventions or prediction of treatment response. Proteomics based on mass spectrometry enables analysis of novel, putative biomarkers. In this study, proteomics was used to analyse in more details extracellular matrix (ECM) proteins and proteins related to ECM signalization which have a well-established role in malignant transformation and invasion of tumor cells.

IGF2 and IGF2R are known biomarkers in cellular metabolism,but their role in oral precancerous lesions, namely oral lichen planus (OLP) as well as in oral squamous cell carcinoma (OSCC) has not been explored so far. The second aim of our study was to analyse IG2F and IGFR2 expression in oral lichen planus and oral squamous cell carcinoma tissues by comparative semiquantitative immunohistochemistry

ELIGIBILITY:
Inclusion Criteria:

* histopathologically confirmed oral lichen planus and oral squamous cell carcinoma
* healthy volunteers referred for alveolotomy

Exclusion Criteria:

* non-consent patients
* previously treated OSCC
* patients under immunosuppressive therapy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A study consisted of 71 consented patients, among which 27 with histologically confirmed diagnosis of oral lichen planus, 23 with oral squamous cell carcinoma and 21 sample of healthy oral mucosa (18 archive samples). Study included 36 male and 35 female patients.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Global proteomic profiling of oral lichen planus and oral squamous cell carcinoma | 2012-2014

SECONDARY OUTCOMES:
evaluation of the Insulin-like growth factor receptor 2 (IGF2R) and IGF2 role in oral lichen planus | 2011-2014

CONTACTS AND LOCATIONS:
Overall Officials: Marinka Mravak-Stipetic, Professor, Principal Investigator — University of Zagreb
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schiller HB, Szekeres A, Binder BR, Stockinger H, Leksa V. Mannose 6-phosphate/insulin-like growth factor 2 receptor limits cell invasion by controlling alphaVbeta3 integrin expression and proteolytic processing of urokinase-type plasminogen activator receptor. Mol Biol Cell. 2009 Feb;20(3):745-56. doi: 10.1091/mbc.e08-06-0569. Epub 2008 Nov 26. PMID 19037107
- [Result] Zavras AI, Pitiphat W, Wu T, Cartsos V, Lam A, Douglass CW, Diehl SR. Insulin-like growth factor II receptor gene-167 genotype increases the risk of oral squamous cell carcinoma in humans. Cancer Res. 2003 Jan 15;63(2):296-7. PMID 12543777
- [Result] Pawar H, Kashyap MK, Sahasrabuddhe NA, Renuse S, Harsha HC, Kumar P, Sharma J, Kandasamy K, Marimuthu A, Nair B, Rajagopalan S, Maharudraiah J, Premalatha CS, Kumar KV, Vijayakumar M, Chaerkady R, Prasad TS, Kumar RV, Kumar RV, Pandey A. Quantitative tissue proteomics of esophageal squamous cell carcinoma for novel biomarker discovery. Cancer Biol Ther. 2011 Sep 15;12(6):510-22. doi: 10.4161/cbt.12.6.16833. Epub 2011 Sep 15. PMID 21743296